CLINICAL TRIAL: NCT07366411
Title: Transcutaneous Auricular Vagus Nerve Stimulation on Functional Mobility in People With Parkinson's Disease
Brief Title: taVNS on Functional Mobility in People With DP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: taVNS_DP
Record Dates: First submitted 2025-12-01; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: PARKINSON DISEASE (Disorder)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcutaneous auricular vagus nerve stimulation (Active Comparator)
  Interventions: Device: Active taVNS
- Sham transcutaneous auricular vagus nerve stimulation (Sham Comparator)
  Interventions: Device: Sham taVNS

INTERVENTIONS:
Device: Active taVNS — taVNS will be applied to the concha in the left auricle of volunteers with the following parameters: 8 trains of 120 seconds of stimulation each at 25 Hz, 300 μs, and 60 seconds of interstimulus interval, with intensity below the pain threshold, totaling 24 minutes of stimulation. The stimulation is combined with physical therapy focused on functional mobility.
  Arms: Active transcutaneous auricular vagus nerve stimulation
Device: Sham taVNS — Physical therapy focusing on functional mobility with sham transcutaneous auricular vagus nerve stimulation.
  Arms: Sham transcutaneous auricular vagus nerve stimulation

SUMMARY:
Parkinson's disease (PD) is characterized by motor impairments such as bradykinesia accompanied by resting tremor and/or rigidity. As PD progresses due to its neurodegenerative nature, complementary strategies must be developed to optimize its effects. Transcutaneous auricular vagus nerve stimulation (taVNS) has emerged as a strategy for controlling the symptoms of the disease. Nevertheless, the efficacy of this approach in managing PD remains to be elucidated. The objective of the present study is to investigate and compare the effects of transcutaneous vagus nerve stimulation (taVNS) and sham taVNS on functional mobility, which is the primary outcome and will be assessed using the Timed Up and Go test. The following tests will be used to evaluate the secondary outcomes: the miniBESTest and the Biodex Balance System (balance), the MDS-UPDRS and the Five-Time Sit-to-Stand Test (motor function), the FOG-Q (freezing of gait), the 10-Meter Walk Test (gait speed), the PGIC (perception of change), and the recording of adverse events. The volunteers will be divided into two groups: one group will receive taVNS in conjunction with physical therapy, while the other group will receive a sham taVNS in conjunction with physical therapy. To assess the effect of therapy, the efficacy of taVNS in enhancing the effects of physical therapy on the functional mobility of people with PD will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of PD provided by a neurologist;
* undergoing regular antiparkinsonian drug treatment (at least three months of regular and stable use);
* aged 40 years or older;
* with a Hoehn & Yahr stage of 2.5 to 4.

Exclusion Criteria:

* other neurological disorders, postural hypotension, vestibular, musculoskeletal, or visual disorders that compromise performance in the proposed tests;
* other osteomyoarticular diseases in the lower limbs that interfere with performance and locomotion;
* Montreal Cognitive Assessment (MoCA) score lower than 21 points;
* previous surgical procedure for PD.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional mobility | Baseline (Day 0), mid-intervention (Day 5), post-intervention (Day 10), 1 month post-intervention (Day 30)
  Functional mobility will be assessed using the Timed Up and Go (TUG) test. In the TUG, the time taken by the volunteer to perform the activity of getting up from a chair, walking, and sitting back down is timed. The test begins with the volunteer sitting in a chair with their back against the backrest; when asked, they stand up, walk three meters at their fastest speed, but safely, turn around, return to the chair, and sit down. Shorter times in performing this test translate into greater functional mobility. Three repetitions of the test will be scored, and for analysis purposes, the average of the repetitions will be used.

SECONDARY OUTCOMES:
Balance | Baseline (Day 0), mid-intervention (Day 5), post-intervention (Day 10), 1 month post-intervention (Day 30).
  Static and dynamic balance will be assessed using the reduced version of the Balance Evaluation System Test (miniBESTest), which aims to evaluate six different balance control mechanisms based on 14 specific activities of daily living. Each activity is scored from 0 (worst performance) to 2 (best performance). Thus, lower scores indicate poorer balance.
Balance | Baseline (Day 0), mid-intervention (Day 5), post-intervention (Day 10), 1 month post-intervention (Day 30)
  The Biodex Balance System (BBS) will be used, which is a mobile platform with levels of instability. In the present study, the postural stability test will be used, starting from level 12 towards level 8. That is, from greater to lesser stability. At the end of the test, the BBS provides three data points: anterior-posterior displacement index (API), medial-lateral displacement index (MLI), and overall stability index (OSI).
Motor function | Baseline (Day 0), mid-intervention (Day 5), post-intervention (Day 10), 1 month post-intervention (Day 30)
  Motor function will be assessed using the Five Times Sit-to-Stand Test (FTSST) and sections II and III of the Movement Disorder Society Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS). In the FTSST, volunteers are asked to stand up and sit down five times as quickly as possible, but safely. Shorter times on this test indicate greater functional mobility. For analysis purposes, the average of three repetitions of this test will be used.
Motor function | Baseline (Day 0), mid-intervention (Day 5), post-intervention (Day 10), 1 month post-intervention (Day 30)
  The MDS-UPDRS is the most widely used clinical assessment tool for characterizing the motor symptoms of PD and for monitoring the progression of these symptoms and the physical disability caused by the disease. The MDS-UPDRS consists of 50 items scored from 0 to 4 each, from best (0) to worst motor performance (4), and is widely accepted for determining the effectiveness of intervention in clinical studies.
Freezing of gait | Baseline (Day 0), mid-intervention (Day 5), post-intervention (Day 10), 1 month post-intervention (Day 30)
  Freezing of gait is assessed using the Freezing of Gait Questionnaire (FOG-Q), which consists of a scale that measures the volunteer's subjective perception of the severity and impact of freezing during gait. The FOG-Q has six items, each scored from 0 to 4, for a total of 24 points. A higher score indicates that gait performance is more affected by freezing.
Speed of gait | Baseline (Day 0), mid-intervention (Day 5), post-intervention (Day 10), 1 month post-intervention (Day 30)
  Walking speed will be assessed using the 10-meter walk test (10MWT), in which the volunteer is instructed to walk down a 10-meter corridor. The test begins with the volunteer standing, and after instruction, they must walk the 10-meter course and stop at the end of it. Two repetitions of the test will be performed, the first with the volunteer walking at their comfortable speed and the second at their fastest speed, but safely.
Patient global impression of change | Post-intervention (Day 10)
  The perception of improvement will be verified through the Patient Global Impression of Change (PGIC). This aims to quantify the volunteer's perception of improvement for the proposed treatment in relation to activities of daily living, disease symptoms, emotions, and quality of life. Volunteers are given seven response options, ranging from "no change or condition worsened" to "much better, with a considerable improvement that made all the difference." This questionnaire will only be administered at the end of the ten sessions.
Adverse events | All days of intervention (up to 10 days)
  Adverse events will be assessed based on the volunteer's report. The most common adverse effects are headache, tingling in the electrode region, burning sensation, and drowsiness. For each sensation, the volunteer will rate its intensity on a Likert scale ranging from 0 (none) to 4 (strong).

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, Phd in neurosciences, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No